CLINICAL TRIAL: NCT03475355
Title: Action Observation Therapy: a Chance for Parkinson's Disease Patients of Improving Mobility Through a Home-based Training
Brief Title: Action Observation Theraphy in Parkinson's Disease
Acronym: ACTIONPARK
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: IRCCS San Camillo, Venezia, Italy (Other)
Collaborators: University of Genova (Other); Università Politecnica delle Marche (Other)
Responsible Party: Principal Investigator, Patrizio Sale, PM&R physician, MD, PhD, University of Padova
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GR-2011-02349761
Record Dates: First submitted 2018-03-16; First posted 2018-03-23 (Actual); Last update posted 2018-03-23 (Actual); Status verified 2018-03

CONDITIONS: Parkinson Disease
Keywords: action observation; parkinson's disease; physical therapy; home-based; neural plasticity; telerehabilitation
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- EG1 (Experimental): Each patient will be instructed to carefully observe the finalized movement of the upper limb of an experimenter seated in front (the experimenter's left hand is right in front of the patient's right hand), without moving or imagining the movement.
  Interventions: Behavioral: Live movement observation (Upper Limbs)
- EG2 (Experimental): Each patient will be instructed to look at a computer screen that is in front of him that will show a daily routine task (actions).
  Interventions: Behavioral: Video Observation (Upper Limbs)
- EG3 (Experimental): Each patient will be instructed to carefully observe the finalized movement performed by an experimenter standing in front of him (the examiner's left leg will be in front of the patient's right leg).
  Interventions: Behavioral: Live Movement Observation (Lowe Limbs)
- EG4 (Experimental): Each patient will be instructed to look at a computer screen that is in front of him that will show a daily routine task (actions).
  Interventions: Behavioral: Video Observation (Lower Limbs)
- CG1 (Active Comparator): Participants will be shown for 3 minutes 5 static images that expose objects, none will represent animals or people.
  The participant's attention will be kept high through a cognitive task. For each CGail patient condition a sequence of images will be presented for 3 minutes, the images will be displayed separately, each for 30 seconds, and then during the last 30 seconds, will be displayed together with an intrusive image (intruder) that the patient will be asked to identify so that his attention span can be controlled in real time. Participants will then be invited to perform movements of the limbs as far as possible for 2 minutes according to a standard sequence that involves articular mobilizations of upper limbs and simulates that performed by the experimental groups.
  Interventions: Behavioral: Static Picture Observation and Upper Limbs Exercise
- CG2 (Active Comparator): Participants will be shown for 3 minutes 5 static images that expose objects, none will represent animals or people.
  The participant's attention will be kept high through a cognitive task. For each CGail patient condition a sequence of images will be presented for 3 minutes, the images will be displayed separately, each for 30 seconds, and then during the last 30 seconds, will be displayed together with an intrusive image (intruder) that the patient will be asked to identify so that his attention span can be controlled in real time. Participants will then be invited to perform movements of the limbs as far as possible for 2 minutes according to a standard sequence that involves articular mobilizations of lower limbs and simulates that performed by the experimental groups.
  Interventions: Behavioral: Static Picture Observation and Lower Limbs Exercise

INTERVENTIONS:
Behavioral: Live movement observation (Upper Limbs) — All participants will be subjected to two 15-minute sessions per day of the Live movement observation of the upper limbs. The activities of the upper limbs will be based on some relevant activities of daily life such as drinking from a glass, combing, opening a box or eating an apple. The tasks will be both unimanual and bimanual.
  Every day, before starting the physical training, the patient will be asked to look carefully at the therapist who shows 20 different daily routine activities (actions) performed with the upper limb.
  Arms: EG1
Behavioral: Video Observation (Upper Limbs) — All participants will be subjected to two 15-minute sessions per day of the video observation of upper limbs movements. The activities of the upper limbs will be based on some relevant activities of daily life such as drinking from a glass, combing, opening a box or eating an apple. The tasks will be both unimanual and bimanual.
  Every day, before starting the physical training, the patient will be asked to carefully watch a video showing 20 different daily routine activities (actions) performed with the upper limb.
  Arms: EG2
Behavioral: Live Movement Observation (Lowe Limbs) — All participants will be subjected to two 15-minute sessions per day of the Live movement observation of the lower limbs. Tasks to avoid freezing will be based on strategies such as touching the thigh, taking side or back steps, counting out loud while walking.
  Every day, before starting the physical training, the patient will be asked to carefully watch the therapist who will show 20 different movement strategies to avoid episodes of freezing the pace (FOG).
  Arms: EG3
Behavioral: Video Observation (Lower Limbs) — All participants will be subjected to two 15-minute sessions per day of the video observation of lower limbs movements. Tasks to avoid freezing will be based on strategies such as touching the thigh, taking side or back steps, counting out loud while walking. Every day, before starting the physical training, the patient will be asked to carefully watch a video that will show 20 different movement strategies to avoid episodes of freezing the pace (FOG).
  Arms: EG4
Behavioral: Static Picture Observation and Upper Limbs Exercise — Participants will watch for 3 minutes 5 static images that expose objects, none will represent animals or people.
  The participant's attention will be kept high through a cognitive task. The patient will be presented a sequence of images for 3 minutes, the images will be displayed separately, each for 30 seconds, and then during the last 30 seconds, they will be displayed together with an intrusive image (intruder) that the patient you will be asked to identify so that your attention span can be controlled in real time. Participants will then be invited to perform limb movements as far as possible for 2 minutes according to a standard sequence involving joint mobilisations of upper limbs, and simulating that performed by the experimental groups.
  Arms: CG1
Behavioral: Static Picture Observation and Lower Limbs Exercise — Participants will watch for 3 minutes 5 static images that expose objects, none will represent animals or people.
  The participant's attention will be kept high through a cognitive task. The patient will be presented a sequence of images for 3 minutes, the images will be displayed separately, each for 30 seconds, and then during the last 30 seconds, they will be displayed together with an intrusive image (intruder) that the patient you will be asked to identify so that your attention span can be controlled in real time. Participants will then be invited to perform limb movements as far as possible for 2 minutes according to a standard sequence involving joint mobilisations of lower limbs, and simulating that performed by the experimental groups.
  Arms: CG2

SUMMARY:
The main objective of this project is to evaluate the effectiveness of Observation of Action (Action Observation, AO) both in increasing the speed of movement of the upper limbs, agility and locomotion, and in improving the activities and quality of life in people with Parkinson's disease (PD) during a 4-6 month follow-up. The second objective is to evaluate the feasibility and effectiveness of a tele-rehabilitation protocol using home-based AO therapy. The telecommunication technology will provide a complete training through a low-cost software run on a touch-screen device, which will show the actions to be imitated several times by people with PD. This project will be the first attempt to implement AO-based treatment at home and, if successful, will be highly translational to clinical practice thanks to the advanced development and broad accessibility of information technology and telecommunications in our country. Furthermore, continuous exercise will reduce the risks of complications and the frequency of hospital admissions, thus reducing costs for the National Health System.

DETAILED DESCRIPTION:
The main objective of this project is to evaluate the effectiveness of Observation of Action (AO) both in increasing the speed of movement of the upper limbs, agility and locomotion, and in improving activities and quality of life in people with Parkinson's disease (PD) during a 4-6 month follow-up. The second objective is to evaluate the feasibility and effectiveness of a tele-rehabilitation protocol using home-based AO therapy. The telecommunication technology will provide a complete training through a low-cost software run on a touch-screen device, which will show the actions to be imitated several times by people with PD. This project will be the first attempt to implement AO-based treatment at home and, if successful, will be highly translational to clinical practice thanks to the advanced development and broad accessibility of information technology and telecommunications in our country. Furthermore, continuous exercise will reduce the risks of complications and the frequency of hospital admissions, thus reducing costs for the National Health System.

Parkinson's disease (PD) should impose a growing social and economic burden on our country. In fact, even with optimal medical management, people with PD experience a worsening of mobility and independence in daily activities, with a consequent reduction in quality of life. In the last ten years there has been a growing demand to consider rehabilitation as an essential adjunct to pharmacological treatment. However, the reference rates for physiotherapy for people with Parkinson's disease have been historically low, both because of poor compliance by patients with the therapies of the movement and because of the scarce availability of physiotherapy services. Action Observation Therapy (AO) has recently been described as an effective strategy in stroke rehabilitation (Sale 2011, 2012), since it can shape the reorganization of the neural circuit, promote neural plasticity and motor learning. . The purpose of this study is to verify the efficacy of AO therapy on PD-related disability and to verify the feasibility of a home-based AO protocol.

The first specific objective of this project is to evaluate the effectiveness of action observation as an additional rehabilitative tool to improve upper limb function in terms of bradykinesia and dexterity and to investigate the stability of treatment effects after 4 / 6 months of follow-up regarding functional improvement and quality of life (QoL). The second specific objective of this project is to evaluate the effectiveness of the observation of the action as an additional rehabilitative tool to improve the balance , gait and, consequently, to reduce falls, and to investigate the stability of treatment effects at 4/6 months of follow-up in terms of functional improvement and quality of life (QoL). The third objective is to evaluate the feasibility and effectiveness of a home telerehabilitation protocol (TR) based on AO therapy to improve dexterity and ambulation in people with Parkinson's disease.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of idiopathic PD according to the UK BRAIN BANK criteria;
* Age between 18 and 80 years;
* Able to walk 25 meters without help or with minimal assistance and sufficient strength to remain standing for at least 20 minutes without assistance for patient report; Stability of drug therapy for Parkinson's disease for at least 4 weeks before the start of the study;
* Mini-Mental State Examination> 25/30;
* HAM-D (Hamilton Depression Scale) <17.

Exclusion Criteria:

* comorbidity with other neurological disorders;
* heart or orthopedic problems;
* Chronic alcohol abuse.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2015-04-22 (Actual); Primary Completion 2018-07-31 (Estimated); Study Completion 2018-10-31 (Estimated)

PRIMARY OUTCOMES:
Box and Block test | 4 weeks
  The Box and Block Test (BBT) measures unilateral gross manual dexterity. It is a quick, simple and inexpensive test. It can be used with a wide range of populations, including clients with stroke.
Nine Hole Peg Test | 4 weeks
  The Nine-Hole Peg Test (9HPT) is used to measure finger dexterity in patients with various neurological diagnoses. Administered by asking the client to take the pegs from a container, one by one, and place them into the holes on the board, as quickly as possible

SECONDARY OUTCOMES:
MDS-UPDRS part II | 4 weeks
  13 items scale focusing on the self-evaluation of the activities of daily life (ADLs) including speech, swallowing, handwriting, dressing, hygiene, falling, salivating, turning in bed, walking, and cutting food. Each subscale now has 0-4 ratings, where 0 = normal, 1 = slight, 2 = mild, 3 = moderate, and 4 = severe.
MDS-UPDRS part III | 4 weeks
  18 items scale based on clinician-scored monitored motor evaluation. Each subscale now has 0-4 ratings, where 0 = normal, 1 = slight, 2 = mild, 3 = moderate, and 4 = severe.
PDQ-39 | 4 weeks
  PDQ-39
  There are 39 questions in the long form Parkinson's Disease Questionnaire, with 8 discrete scales: mobility (10 items); activities of daily living (6 items); emotional well-being (6 items); stigma (4 items); social support (3 items); cognitions (4 items); communication (3 items); bodily discomfort (3 items). Patients are asked to think about their health and general well-being and to consider how often in the last month they have experienced certain events (e.g. difficulty walking 100 yards). Patients are asked to indicate the frequency of each event by selecting one of 5 options (likert Scale): never/occasionally/sometimes/often/always or cannot do at all.
Small Coin Rotation Test | 4 weeks
  The coin rotation task (CRT) is a simple, convenient, and cost-effective measure of psychomotor processing speed. In the CRT, participants rotate a coin through serial 180-degree turns using the thumb, index, and middle fingers for 10 seconds.
Small Lock Rotation Test | 4 weeks
Clinical Global Impression Scale | 4 weeks
  The Clinical Global Impression (CGI) rating scales are measures of symptom severity, treatment response and the efficacy of treatments in treatment studies
3D Movement Analysis | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Infarinato, PhD, Study Director — IRCCS San Raffaele; Patrizio Sale, PhD, Principal Investigator — Univesity of Padua
Locations (1):
- IRCCS San Camillo Hospital, Venezia, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Franceschini M, Ceravolo MG, Agosti M, Cavallini P, Bonassi S, Dall'Armi V, Massucci M, Schifini F, Sale P. Clinical relevance of action observation in upper-limb stroke rehabilitation: a possible role in recovery of functional dexterity. A randomized clinical trial. Neurorehabil Neural Repair. 2012 Jun;26(5):456-62. doi: 10.1177/1545968311427406. Epub 2012 Jan 10. PMID 22235059
- [Background] Pelosin E, Bove M, Ruggeri P, Avanzino L, Abbruzzese G. Reduction of bradykinesia of finger movements by a single session of action observation in Parkinson disease. Neurorehabil Neural Repair. 2013 Jul-Aug;27(6):552-60. doi: 10.1177/1545968312471905. Epub 2013 Feb 7. PMID 23392919
- [Background] Cross ES, Liepelt R, Hamilton AF, Parkinson J, Ramsey R, Stadler W, Prinz W. Robotic movement preferentially engages the action observation network. Hum Brain Mapp. 2012 Sep;33(9):2238-54. doi: 10.1002/hbm.21361. Epub 2011 Sep 6. PMID 21898675
- [Background] Alegre M, Guridi J, Artieda J. The mirror system, theory of mind and Parkinson's disease. J Neurol Sci. 2011 Nov 15;310(1-2):194-6. doi: 10.1016/j.jns.2011.07.030. Epub 2011 Aug 11. PMID 21839480
- [Background] Buccino G, Gatti R, Giusti MC, Negrotti A, Rossi A, Calzetti S, Cappa SF. Action observation treatment improves autonomy in daily activities in Parkinson's disease patients: results from a pilot study. Mov Disord. 2011 Aug 15;26(10):1963-4. doi: 10.1002/mds.23745. Epub 2011 May 5. No abstract available. PMID 21547952
- [Background] Pelosin E, Avanzino L, Bove M, Stramesi P, Nieuwboer A, Abbruzzese G. Action observation improves freezing of gait in patients with Parkinson's disease. Neurorehabil Neural Repair. 2010 Oct;24(8):746-52. doi: 10.1177/1545968310368685. Epub 2010 May 7. PMID 20453155
- [Background] Sale P, Franceschini M. Action observation and mirror neuron network: a tool for motor stroke rehabilitation. Eur J Phys Rehabil Med. 2012 Jun;48(2):313-8. Epub 2012 Apr 20. PMID 22522432
- [Background] Alegre M, Rodriguez-Oroz MC, Valencia M, Perez-Alcazar M, Guridi J, Iriarte J, Obeso JA, Artieda J. Changes in subthalamic activity during movement observation in Parkinson's disease: is the mirror system mirrored in the basal ganglia? Clin Neurophysiol. 2010 Mar;121(3):414-25. doi: 10.1016/j.clinph.2009.11.013. Epub 2009 Dec 16. PMID 20006544
- [Background] Franceschini M, Agosti M, Cantagallo A, Sale P, Mancuso M, Buccino G. Mirror neurons: action observation treatment as a tool in stroke rehabilitation. Eur J Phys Rehabil Med. 2010 Dec;46(4):517-23. Epub 2010 Apr 23. PMID 20414184